CLINICAL TRIAL: NCT06483724
Title: Comparison Between Cervical Tourniquet and Uterine Artery Ligation Prior to the Segmental Resection Approach in Patients With Placenta Accreta Spectrum: A Prospective Interventional Study
Brief Title: Comparison Between Cervical Tourniquet and Uterine Artery Ligation Prior to Segmental Resection Approach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Mohamed Abdel Ghfar, lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Placenta Accreta Spectrum
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (n = 41) cervical tourniquet (Experimental): in group 1 the investigators using a sterile Foley catheter (Ch 16/18 French) down to the lowest point and secures it "en bloc" around the cervix at the level of the uterosacral ligaments, approximately 3-4 cm below the incision. Then, tighten and fix .
  Interventions: Procedure: cervical tourniquet
- Group 2 (n=41) uterine artery ligation (Experimental): in group 2the investigators ligated the uterine vessels in a continuous manner at the level of the utero-vesical fold on each side.
  Interventions: Procedure: uterine artery ligation

INTERVENTIONS:
Procedure: cervical tourniquet — After opening the abdominal wall, To reduce bleeding during PAS, make the uterine incision above the placenta's intrauterine borders .
  2-investigators extract the uterus from the abdomen 3-An assistant slides a sterile Foley catheter (Ch 16/18 French) down to the lowest point and secures it "en bloc" around the cervix 4-The bladder peritoneum is isolated from the uterus 5-To remove myometrial tissue, leave a margin of at least 2 cm superior to the cervical internal ostium using electrocautery or scissors .
  Arms: Group 1 (n = 41) cervical tourniquet
Procedure: uterine artery ligation — After opening the abdominal wall, To reduce bleeding during PAS, make the uterine incision above the placenta's intrauterine borders .
  2-investigators extract the uterus from the abdomen 3-The bladder peritoneum is isolated from the uterus 4-The uterine vessels were ligated in continuity at the level of the utero-vesical fold on each side 5-To remove myometrial tissue, leave a margin of at least 2 cm superior to the cervical internal ostium using electrocautery or scissors .
  Arms: Group 2 (n=41) uterine artery ligation

SUMMARY:
The study will compare a modified surgical approach for preserving fertility and minimizing hemorrhage in morbidly adherent placenta during cesarean section with a cervical tourniquet against uterine artery ligation.

DETAILED DESCRIPTION:
Study Design and Setting This was prospective interventional study that comprised the medical data of 82 pregnant women with placenta accreta who had caesarean section. . This study will be carried out In the Department of Obstetrics and Gynecology, Minia Maternity University Hospital (MMUH) .

after being approved by the local ethical Committee; If placenta accreta was clinically verified preoperatively, all parturients were informed of the option of a hysterectomy. After receiving written, formal consent . After receiving documented formal consent. The study included all patients who had a scheduled cesarean procedure for placenta accreta. Obstetrical imaging either verified or strongly suspected the diagnosis. During the prenatal period, a senior sonographer evaluated all patients using ultrasonography and color Doppler technology. An ultrasonographic assessment was done. Each patient was evaluated for retroplacental sonolucent zones, vascular lacunas, myometrial thinning, bladder line disruption, and exophytic masses . The Color Doppler scan evaluated placental lacunar flow, hypervascularity in the vesicouterine interface, and continuous retroplacental venous complex structures. A 3D Doppler scan was used to assess hypervascularity of the uterine serosa and bladder interphase, as well as uneven intraplacental vascularization

Assessment :

To assess the effectiveness of the proposed management strategy, participants were separated into two groups. In Group 1 (n = 41), a cervical tourniquet was used systematically. In Group 2 (n=41), uterine artery ligation was performed prior to segmental resection for uterine preservation surgery

Surgical scenarios :

Across both groups: Ultrasonographic data determine whether an abdominal incision should be performed with a Pfannensteil or a vertical midline incision from under the umbilicus to above the pubic symphysis.

1. in group 1 After opening the abdominal wall, To reduce bleeding during PAS, make the uterine incision above the placenta's intrauterine borders. Before making the incision, an ultrasound check is recommended to find the uterine opening. Based on our assumptions, following the delivery of the fetus
2. investigators was extract the uterus from the abdomen by gently grasp the fundus of the uterus and pull up and forward. Release uterine appendages on both sides by shifting the uterus to the right and left.
3. An assistant slides a sterile Foley catheter (Ch 16/18 French) down to the lowest point and secures it "en bloc" around the cervix at the level of the uterosacral ligaments, approximately 3-4 cm below the incision. Then, tighten and fix it.
4. The bladder peritoneum is isolated from the uterus through complex coagulation of perforating vascular systems . This step of surgery is crucial for the rest of the treatment. Due to the fragile and unpredictable nature of the vascular network, it is important to exercise caution. The bladder peritoneum is demarcated until the cervical internal ostium. To accomplish this procedure, an assistant places a finger on the anterior fornix of the vagina to create a reference point and assure full separation.
5. To remove myometrial tissue, leave a margin of at least 2 cm superior to the cervical internal ostium using electrocautery or scissors.
6. The tourniquet approach achieves hemostasis, giving the operator time to assess the uterus's preservation potential.
7. To assess active bleeding, the tourniquet can be removed.
8. Suturing on the uterine pouches by suturing on the Uterine pouches is repaired by bringing the edges together with running sutures or using the internal os of the cervix as a natural tamponade helps produce hemostasis in the placental bed and adjacent areas.
9. This approach provides time to prepare for a blood transfusion or seek assistance. The tourniquet approach can be utilized as both a primary therapy strategy for PAS and a follow-up after placental removal and bleeding.

In another group : the same steps in group 1 in steps 1, 2 and 3 4- The bladder peritoneum is isolated from the uterus 5 - The uterine vessels were ligated in continuity at the level of the utero-vesical fold on each side.

6- the same steps in group 1 in steps 5,6, 7and 8

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed sonographically to have placenta accreta spectrum .
* Pregnancy is singleton and fetus is alive.
* Elective caesarean section done from 36 gestational weeks

Exclusion Criteria:

* Patients requesting hysterectomy
* Coexisting uterine pathology such as fibroids or gynaecological malignancies
* Patients with bleeding diathesis.
* Morbid obesity of BMI >40.
* Patients having labour pains or vaginal bleeding before scheduled intervention

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
operation time | intraoperative
  recording total time of the surgery
repair time | intraoperative
  recording length of defect repair from placental separation until uterine wall closure
Estimated blood loss | intraoperative
  recording amount of blood loss
packed red blood cells transfusion | intraoperative until 24 hours after surgery
  recording amount of red blood cell transfused
fresh frozen plasma (FFP) transfusion | intraoperative until 24 hours postoperative
  recording amount of FFP transfusion
Number of Participants who had Bladder injuries | intraoperative until 2 weeks post operative
  Number of Participants who had Bladder injuries
Number of Participants who had ureteral injuries | intraoperative until 2 weeks post operative
  Number of Participants who had ureteral injuries
Number of Participants who had bowel injury | intraoperative until 2 weeks post operative
  Number of Participants who had bowel injury
surgical site infection | 24 hours until 1 month after surgery
  record the presence of wound infection
urine output | intraoperative
  recording amount of urine output
internal iliac artery ligation | intraoperative
  recording if the internal iliac artery ligated whether it was unilateral or bilateral
pre-operative hemoglobin | preoperative
  recording amount of hemoglobin
post-operative hemoglobin | postoperative within 6 hours from surgery
  recording amount of hemoglobin
hospital stay | postoperative until 10 days after surgery
  recording duration of hospital stay after surgery
ICU admission | immediate postoperative until 5 days after surgery
  recording the number of patients admitted to the ICU
HDU high dependency unit admission | postoperative until 10 days after surgery
  recording the number of patients admitted to high dependency unit
surgical diagnosis | intraoperative
  strategy to preserving the uterus when managing placenta accreta versus hysterectomy

IPD SHARING:
Plan to Share IPD: No